CLINICAL TRIAL: NCT04037072
Title: GI-108: Randomized Controlled Double-Blinded Trial Assessing the Efficacy of Topical Mitomycin C for Complex Benign Esophageal Anastomotic Strictures
Brief Title: Efficacy of Topical Mitomycin C for Complex Benign Esophageal Anastomotic Strictures
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not approved for Fox Chase Cancer Center's Research Review Committee (RRC)
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-1022
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Stenosis; Anastomotic Stenosis
Keywords: Complex
MeSH Terms: conditions — Esophageal Stenosis | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mitomycin C (Experimental): Cotton swab or strip of 2x2 cotton gauze soaked with 0.4mg/mL Mitomycin C
  Interventions: Drug: Mitomycin C
- Control (Placebo Comparator): Cotton swab or strip of 2x2 cotton gauze soaked with Normal saline
  Interventions: Other: Control

INTERVENTIONS:
Drug: Mitomycin C — Topical application of Mytomycin C (MMC)
  Other Names: MMC
  Arms: Mitomycin C
Other: Control — Topical application of Normal Saline
  Other Names: NS
  Arms: Control

SUMMARY:
This study evaluates Mitomycin C as treatment for dysphagia in adult subjects with documented complex esophageal anastomotic strictures. Patients will be randomized in a double-blinded fashion to topical application of normal saline (NS) or Mitomycin C (MMC) at the time of time of index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Patients must have symptomatic (dysphagia ≥2), treatment naïve complex esophageal anastomotic stricture (length >2 cm or diameter ≤9mm).
* Age ≥ 18
* Esophago-gastro or esophago-jejunal anastomosis with or without having undergone neoadjuvant or adjuvant radio-chemotherapy
* Any patient taking antiplatelet agents such as Plavix, Effient, Brilinta, Aggrenox must be able to hold the drugs 5 days prior to dilation and may resume 3 days after the dilation.
* Any patient on vitamin K antagonists such as warfarin must be able to hold the drugs 5 days prior to dilation and may resume 3 days after the dilation. INR should be checked for such patients at least 24 hours before dilation and it must be < 1.5
* Patients taking direct thrombin inhibitors such as Pradaxa, Angiomax must be able to hold the drugs 5 days prior to dilation and may resume 3 days after the dilation
* Patients taking Factor Xa inhibitors must be able to hold the drugs 2 days prior to dilation and may resume 3 days after dilation
* Patients taking GIIB/IIIA inhibitors must be able to hold the drugs1 day prior to dilation and resume 3 days after the dilation.
* Patients taking unfractionated heparin must be able to hold the drug 6 hours before dilation and low molecular weight heparin must be held 24 hours before dilation. Unfractionated heparin may resume immediately after the dilation while low molecular weight heparin may resume 3 days after dilation

Exclusion Criteria:

* Patients with malignant strictures
* Patients with non-complex benign strictures.
* Patients with anastomosis creation within ≤ 2 weeks
* Patients with suspected gastrointestinal perforation or leak that could result in extraluminal extravasation of Mitomycin C
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding. Refer to section 4.4 for further detail.
* Patients receiving systemic chemotherapy during the treatment of esophageal stricture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of dysphagia ≥ grade 1 after the dilation procedure | 6 months
  Prevalence of dysphagia grade ≥1 in MMC Vs normal saline treated patients until 6 months after the first follow-up.

SECONDARY OUTCOMES:
Number of procedures needed to reach dilation goal | 30 days
  calculated from the first treatment procedure until the last one and will be compared between the experimental and the control arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States